CLINICAL TRIAL: NCT01176019
Title: An Interactive Informed Consent and Education Program for Pregnant Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: ArchieMD (Unknown)
Responsible Party: Principal Investigator, William Grobman, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NIH-291
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy; Down Syndrome
Keywords: Amniocentesis; Chorionic Villus Sampling; First trimester screening; Down syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Diagnosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interactive Video (Experimental): In addition to standard care, the experimental arm will receive an interactive video designed to inform and educate patients about the choices that exist concerning prenatal screening and diagnosis.
  Interventions: Device: Information about Prenatal Screening and Diagnosis
- Control (No Intervention): A control arm will receive standard care, which is the opportunity to meet with a genetic counselor.

INTERVENTIONS:
Device: Information about Prenatal Screening and Diagnosis — 15-20 minute interactive video about prenatal screening and diagnosis given on day of recruitment.
  Arms: Interactive Video

SUMMARY:
The purpose of this study is to determine whether an interactive education program for prenatal testing is effective in improving pregnant women's understanding of and expectations towards prenatal screening and diagnosis.

DETAILED DESCRIPTION:
Women face a variety of medical decisions during pregnancy and childbirth. While there are extensive educational resources for pregnant women, modern medicine presents decisions that many women are poorly equipped to make. Issues such as prenatal screening and mode of birth after a cesarean delivery require a significant degree of patient education to enable a truly informed medical decision. Studies have shown that women have a poor understanding of screening for birth defects and mode of birth after a cesarean delivery. Women with a low level of education or poor health literacy are significantly more likely to demonstrate inadequate understanding of prenatal screening. ArchieMD, Inc. has developed a comprehensive interactive medical simulation environment which has the potential to visually convey complex information to patients to improve understanding of medical procedures and educate patients on the consequences of their behavior. We hypothesize that such an interactive medical simulation patient education program can improve patient understanding allowing pregnant women to make informed decisions. In Phase I, we will prototype an interactive patient education program for prenatal screening and amniocentesis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman (6-26 weeks gestation)
* Over 18 years of age

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Difference in understanding/knowledge gain as compared to control | Post-test and 2 week follow-up
  Open-ended and T/F questionnaire designed to determine if the ArchieMD Interactive Informed Consent and Education Program for Pregnant Women improves understanding and expectations of prenatal screening and diagnostic tests in a group of pregnant women patients.

SECONDARY OUTCOMES:
eHEALS | Post-test
  The eHEALS is a self-report tool that can be administered by a health professional and is based on an individual's perception of her or his own skills and knowledge within each measured domain. The instrument is designed to provide a general estimate of consumer eHealth-related skills that can be used to inform clinical decision making and health promotion planning with individuals or specific populations.
Attitudes towards/satisfaction with interactive video | Post-test
  Multiple-choice questionnaire designed to determine if the ArchieMD Interactive Informed Consent and Education Program for Pregnant Women enhances satisfaction with and attitudes toward the patient education process.
REALM | Post-test
  The REALM (Rapid Estimate of Adult Health Literacy in Medicine) is a word recognition test designed to provide a valid and quick assessment of participant health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Grobman, M.D., M.B.A, Principal Investigator — Northwestern University; Michael Wolf, Ph.D, M.P.H, Principal Investigator — Northwestern University; Robert Levine, M.D., Principal Investigator — ArchieMD, Inc.
Locations (2):
- United States (2):
  - Northwestern Memorial Faculty Foundation (NMFF), Chicago, Illinois
  - Northwestern Memorial Hospital (NMH), Chicago, Illinois